CLINICAL TRIAL: NCT00649883
Title: A Phase II, Observer-Blind, Randomized, Multi-center Study to Evaluate the Safety and Immunogenicity of Two 0.25 mL or 0.5 mL Doses of Investigational Vaccine and Active Influenza Vaccine in Healthy Children Aged 6 to <60 Months
Brief Title: Safety and Immunogenicity of Two 0.25 mL or 0.5 mL Doses of Two Different Influenza Vaccines in Healthy Children Aged 6 to <60 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V70P6
Record Dates: First submitted 2008-03-25; First posted 2008-04-01 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: Influenza; vaccine; children
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Influenza Trivalent Inactivated vaccines Novartis
- 2 (Active Comparator)
  Interventions: Biological: Influenza Trivalent Inactivated vaccines

INTERVENTIONS:
Biological: Influenza Trivalent Inactivated vaccines Novartis — Children 6 to <36 months of age will receive two 0.25 mL doses, and children 36 to <60 months of age will receive two 0.5 mL doses of investigational influenza vaccine, administered four weeks apart intramuscularly (IM) in the deltoid muscle preferably of the non-dominant arm.
  Arms: 1
Biological: Influenza Trivalent Inactivated vaccines — Children 6 to <36 months of age will receive two 0.25 mL doses, and children 36 to <60 months of age will receive two 0.5 mL doses of active control influenza vaccine, administered four weeks apart intramuscularly (IM) in the deltoid muscle preferably of the non-dominant arm.
  Arms: 2

SUMMARY:
This a multicenter phase II trial will evaluate safety and immunogenicity of two 0.25 mL or 0.5 mL doses of investigational influenza vaccine and active control influenza vaccine in healthy children aged 6 to <60 months.

ELIGIBILITY:
Inclusion Criteria:

* Children of 6 to <60 months of age, whose parents/legal guardians have given written informed consent prior to study entry.
* In good health as determined by: medical history, physical examination, clinical judgment of the investigator.
* Able to comply with all study procedure

Exclusion Criteria:

* Any serious disease, such as: cancer,autoimmune disease (including rheumatoid arthritis), diabetes mellitus, chronic pulmonary disease, acute or progressive hepatic and renal disease, acute or progressive neurological or neuromuscular disease;
* History of any anaphylaxis or serious reaction following administration of vaccine, or hypersensitivity to eggs, egg protein, chicken feathers, influenza viral protein, or any other vaccine component, chemically related substance, or component of the potential packaging materials;
* Known or suspected impairment/alteration of immune function, including: immunosuppressive therapy, cancer chemotherapy, receipt of immunostimulants within 60 days prior to Visit 1, receipt of parenteral immunoglobulin known HIV infection or HIV-related disease;
* Bleeding diathesis;
* Surgery planned during the study period;
* Receipt of another investigational agent within 90 days
* Laboratory-confirmed influenza disease within 6 months prior to Visit 1;
* Ever received two doses of an influenza vaccine before the study
* Receipt of an influenza vaccine within 6 months prior to Visit 1;
* Experienced a temperature 38.0°C within 3 days prior to Visit 1

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of one and two doses of investigational vaccines or active control influenza vaccine in unprimed healthy children aged 6 months to <36 months. | 211 days

SECONDARY OUTCOMES:
To evaluate the immunogenicity of two doses of investigational influenza vaccine or active control influenza vaccines, as measured by HI assay in children aged 36 to <60 months. | 211 days

CONTACTS AND LOCATIONS:
Locations (5):
- Guatemala (5):
  - Centro Clínico La Quinta, Guatemala City, Guatemala City
  - Clínicas Dr. Rafael Montiel, Guatemala City, Guatemala City
  - Dr. Carlos Fernando Grazioso Aragón, Guatemala City, Guatemala City
  - Fundación Pediátrica Guatemalteca, Guatemala City, Guatemala City
  - Hospital Infantil de Infectologia y rehabilitacion, Guatemala City, Guatemala City